CLINICAL TRIAL: NCT04335916
Title: Multicenter Assessment of Pre-Electroconvulsive Therapy (ECT) Evaluation and ECT Application
Brief Title: Survey on Pre-ECT Evaluation and ECT Application
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinički Bolnički Centar Zagreb (Other)
Responsible Party: Sponsor
Other Study IDs: KBC Zagreb
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Depression; Catatonia; Schizophrenia; Schizoaffective Disorder; Suicidal Intention; Malignant Neuroleptic
Keywords: Electroconvulsive therapy; Pre-ECT evaluation
MeSH Terms: conditions — Depression; Catatonia; Schizophrenia; Psychotic Disorders; Neuroleptic Malignant Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify specifics of pre-ECT assessments and ECT application in European psychiatric services. We will engage European centres that provide ECT for psychiatric patients and for psychiatric indications. It could bring better insights on current standards and possibly give some further improvements in the field of European ECT practices.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is an extremely important therapeutic method in the treatment of certain psychiatric conditions. Its' effect has been demonstrated in many clinical trials, and the indications for the use of ECT are clearly defined. Thus, the absolute indications for the use of ECT are catatonia and malignant neuroleptic syndrome, while the relative indications for ECT are therapy-resistant schizophrenia, depression and chronic suicidality. When the lead psychiatrist sets an indication for the use of ECT, pre-ECT evaluation is conducted. Although the pre-evaluation aims to assess the psychophysical condition of the patient and to determine the potential risks and possible side effects of such therapy, no clear algorithm of procedures is specified. There is no data on clear guidelines for the necessary processing prior to the application of ECT, both at national levels and globally. The assessment recommendations, however, are very broad, and most of them are focused on the ethical issues of applying ECT. The standardized pre-ECT evaluation would provide physicians and patients a systematic and evidence-based risk assessment and presumption of adverse reaction profiles.

ELIGIBILITY:
Inclusion Criteria:

* departments that provide pre-ECT assessment
* departments that provide ECT application
* departments that provide both pre-ECT assessment and ECT application

Exclusion Criteria:

* departments that used to provide either pre-ECT assessment or ECT application
* departments that refer patients for ECT but don't provide pre-ECT assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Departments that provide pre-ECT assessment, ECT application or both in Europe
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
pre-ECT evaluation data | Baseline
  Data on pre-ECT evaluation collected with specially designed survey for this research.
  Pre-ECT evaluation treatment includes are there written or agreed indications, inclusion and exclusion criteria and pre-ECT evaluation, the common neuropsychiatric and somatic evaluation for ECT candidate.
ECT administration data | Baseline
  Data on ECT application collected with specially designed survey for this research. The survey examines the most common methods of applying ECT, provided education and the necessary legal and ethical codes.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinički Bolnički Centar Zagreb, Zagreb, City of Zagreb, Croatia

REFERENCES:
- [Derived] Medved S, Zaja N, Gazdag G, Lengvenyte A, Morkl S, Mucci F, Ristic I, Jerotic S, Regente JF, Ivanovic I, Purisic A, Sasvary F, Sivasanker V, Ziblak A, Lookene M, Sienaert P, Szczegielniak A, Trancik P, Becirovic E, Koutsomitros T, Grech G, Tapoi C, Radmanovic B, Strohle A, Bajs Janovic M, Sartorius N. Preliminary Assessment of Pre-Electroconvulsive Therapy Evaluation Practices in European Countries: The Need for Guidelines. J ECT. 2022 Dec 1;38(4):230-237. doi: 10.1097/YCT.0000000000000854. Epub 2022 Apr 23. PMID 35462388